CLINICAL TRIAL: NCT06246214
Title: Innovations in Biological Rhythms in the Context of Mental Health: Effectiveness of New Technologies and Exposure to Different Lighting Patterns in Women During the Postpartum Period
Brief Title: From Prevention to Treatment: How Biological Rhythms Can Maintain Perinatal Mental Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-0584
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Depression, Postpartum; Anxiety State
MeSH Terms: conditions — Depression, Postpartum; Anxiety Disorders | interventions — Phototherapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- BlueLT (Active Comparator): Participants with depressive and/or anxiety symptoms that will receive the interventional light (BlueLT)
  Interventions: Device: Blue Light Therapy
- ControlLT (Sham Comparator): Participants with depressive and/or anxiety symptoms that will receive the placebo light (ControlLT)
  Interventions: Device: ControlLT
- Healthy control (No Intervention): Participants without depressive and/or anxiety symptoms

INTERVENTIONS:
Device: Blue Light Therapy — The BlueLT device is equipped with a narrow band short wavelength Light Emitting Diode (LED) - wavelength peak(λp) of ~470 nm (blue).
  Arms: BlueLT
Device: ControlLT — The ControlLT (placebo) device is equipped with a dim long-wavelength enriched LED.
  Arms: ControlLT

SUMMARY:
Depression and anxiety are significant public health issues during pregnancy and the postnatal period, particularly affecting those in developing countries. Disruptions in biological rhythms, sleep problems, and low exposure to daylight are associated with a higher risk of these mental health issues. The perinatal period poses unique challenges to the temporal program, with evidence indicating that sleep disturbances significantly increase the risk of postnatal depression. A Randomised Clinical Trial (RCT) is being conducted to assess the effectiveness of Blue Light Therapy (BlueLT) in treating depressive and anxiety symptoms during the postpartum. The RCT will also investigate the alignment of rest-activity and internal body time as mediating factors. This study will focus on various chronobiological factors, including rest-activity rhythms, light exposure levels, temperature rhythms, sleep duration and phase, social jetlag, and BodyTime (assessed through a single blood sample). The goal is to recruit 50 women with postpartum depression, with 25 in the BlueLT intervention group and 25 in the ControlLT placebo group, alongside 100 healthy controls. The BlueLT device uses a short-wavelength LED lamp mainly composed by a wavelength peak on blue spectrum, while the ControlLT device has a dim long-wavelength LED. A Healthy Control group will also be included to account for changes unrelated to depression diagnosis or placebo/treatment effects. Exclusion criteria involve a history of major depressive or anxiety disorder, current psychotic disorder, night shift work, active suicidal thoughts, unstable medical conditions interfering with data collection, and newborns with severe health conditions. The study aims to evaluate the impact of BlueLT on postpartum depression and understand the role of chronobiological factors in the health/disease process.

DETAILED DESCRIPTION:
Depression and anxiety during pregnancy and the postnatal period are major public health concerns, particularly in low and middle-income settings. Alterations in biological rhythms, sleep disturbances, and reduced exposure to daylight have been associated with increased risk for these conditions. The perinatal period represents a unique model of circadian misalignment vulnerability, driven by specific challenges to the temporal organization of physiological and behavioral rhythms. Prior evidence indicates that increased sleep onset latency and sleep deficits elevate the risk of postnatal depression, with sleep disturbances being among the most prominent risk factors and associated with up to a four-fold increase in depression risk.

Emerging findings suggest that changes in circadian health indicators, including sleep patterns, rest-activity rhythms, and light exposure, play a significant role in mood regulation during the peripartum period. Chronobiological interventions may therefore represent promising strategies for both prevention and treatment.

This Randomised Clinical Trial (RCT) aims to evaluate the effectiveness of Blue Light Therapy (BlueLT) for reducing depressive symptoms in women with postpartum depression and to assess whether alignment between rest-activity rhythms and internal body time mediates treatment effects. Chronobiological measures will include rest-activity rhythms, light exposure patterns, temperature rhythms, sleep duration and timing, social jetlag, and the BodyTime assay (single blood sample).

Participants with postpartum depression will be randomly assigned to either the BlueLT intervention or placebo light therapy (ControlLT). The BlueLT device delivers short-wavelength, narrow-band LED light (λp ~470 nm), while the ControlLT device emits dim, long-wavelength-enriched light. All participants in both groups will use the assigned light device for 30 minutes each day before 16:00 (4 p.m.) for 30 consecutive days.

The trial will enroll 50 women with postpartum depression (25 in the BlueLT group and 25 in the ControlLT group) and an additional 100 healthy postpartum controls from the same cohort. This healthy control group will serve as a comparator for circadian changes unrelated to depressive symptoms or treatment/placebo effects, acknowledging that pregnancy and postpartum adaptations may independently affect circadian phase relationships.

Exclusion criteria include: history of major depressive or anxiety disorder; current psychotic disorder; night-shift work; active suicidal ideation or psychotic symptoms; unstable medical conditions interfering with actigraphy; and newborns with severe health conditions.

ELIGIBILITY:
Inclusion Criteria:

* 4-6 weeks postpartum;
* Postnatal depression confirmed through Edinburgh Postnatal Depression Scale (EPDS) > 10;
* Mini-International Neuropsychiatric Interview (M.I.N.I.) positive for current depressive episode.

Exclusion Criteria:

* Active suicidal ideation;
* Psychotic symptoms;
* Unstable general medical conditions that interfere with the acquisition of actigraphy;
* Newborn with severe health conditions (hospitalization, care in the neonatal ICU).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-01-04 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms | From enrollment to the end of treatment at 4 weeks
  The EDPS was developed to identify women who may have postpartum depression. This scale consists of 10 short statements. The participant checks off one of four possible answers that is closest to how she has felt during the past week. Responses are scored 0, 1, 2 and 3 based on the seriousness of the symptom. Items 3, 5 to 10 are reverse scored (i.e., 3, 2, 1, and 0). The total score is found by adding together the scores for each of the 10 items. A total score higher than 10 indicate the presence of depressive symptoms. A reduction in depressive symptoms clinically significant (outcome measure) will consist in a minimum difference of 4 points on the EPDS.
Anxiety symptoms | From enrollment to the end of treatment at 4 weeks
  The General Anxiety Disorder 7-item scale (GAD-7) is one of the tools used to screen for anxiety or to measure its severity. Total score is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." Ranging from 0 to 21, the following threshold were previously proposed: 0-4 (minimal anxiety); 5-9 (mild anxiety); 10-14 (moderate anxiety); 15-21 (severe anxiety). A reduction in anxiety symptoms clinically significant (outcome measure) will consist in a minimum difference of 4 points on the GAD-7.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Paz L Hidalgo, Principal Investigator — +555133596339
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tonon AC, Constantino DB, Amando GR, Abreu AC, Francisco AP, de Oliveira MAB, Pilz LK, Xavier NB, Rohrsetzer F, Souza L, Piccin J, Caye A, Petresco S, Manfro PH, Pereira R, Martini T, Kohrt BA, Fisher HL, Mondelli V, Kieling C, Hidalgo MPL. Sleep disturbances, circadian activity, and nocturnal light exposure characterize high risk for and current depression in adolescence. Sleep. 2022 Jul 11;45(7):zsac104. doi: 10.1093/sleep/zsac104. PMID 35522984
- [Background] Roenneberg T, Foster RG, Klerman EB. The circadian system, sleep, and the health/disease balance: a conceptual review. J Sleep Res. 2022 Aug;31(4):e13621. doi: 10.1111/jsr.13621. Epub 2022 Jun 7. PMID 35670313
- [Background] Hidalgo MP, Caumo W, Posser M, Coccaro SB, Camozzato AL, Chaves ML. Relationship between depressive mood and chronotype in healthy subjects. Psychiatry Clin Neurosci. 2009 Jun;63(3):283-90. doi: 10.1111/j.1440-1819.2009.01965.x. PMID 19566758
- [Background] Xavier NB, Abreu ACVO, Amando GR, Steibel EG, Pilz LK, Freitas JJ, da Silveira Cruz-Machado S, Markus RP, Frey BN, Hidalgo MP. Chronobiological parameters as predictors of early treatment response in major depression. J Affect Disord. 2023 Feb 15;323:679-688. doi: 10.1016/j.jad.2022.12.002. Epub 2022 Dec 5. PMID 36481230
- [Background] Kramer A, Lange T, Spies C, Finger AM, Berg D, Oster H. Foundations of circadian medicine. PLoS Biol. 2022 Mar 24;20(3):e3001567. doi: 10.1371/journal.pbio.3001567. eCollection 2022 Mar. PMID 35324893
- [Background] Krawczak EM, Minuzzi L, Simpson W, Hidalgo MP, Frey BN. Sleep, daily activity rhythms and postpartum mood: A longitudinal study across the perinatal period. Chronobiol Int. 2016;33(7):791-801. doi: 10.3109/07420528.2016.1167077. Epub 2016 Apr 20. PMID 27097327
- [Background] Slyepchenko A, Minuzzi L, Reilly JP, Frey BN. Longitudinal Changes in Sleep, Biological Rhythms, and Light Exposure From Late Pregnancy to Postpartum and Their Impact on Peripartum Mood and Anxiety. J Clin Psychiatry. 2022 Jan 18;83(2):21m13991. doi: 10.4088/JCP.21m13991. PMID 35044728
- [Background] Pilz LK, Carissimi A, Francisco AP, Oliveira MAB, Slyepchenko A, Epifano K, Garay LLS, Fabris RC, Scop M, Streiner DL, Hidalgo MP, Frey BN. Prospective Assessment of Daily Patterns of Mood-Related Symptoms. Front Psychiatry. 2018 Aug 21;9:370. doi: 10.3389/fpsyt.2018.00370. eCollection 2018. PMID 30186188
- [Background] Pilz LK, Keller LK, Lenssen D, Roenneberg T. Time to rethink sleep quality: PSQI scores reflect sleep quality on workdays. Sleep. 2018 May 1;41(5). doi: 10.1093/sleep/zsy029. PMID 29420828
- [Background] Pilz LK, Carissimi A, Oliveira MAB, Francisco AP, Fabris RC, Medeiros MS, Scop M, Frey BN, Adan A, Hidalgo MP. Rhythmicity of Mood Symptoms in Individuals at Risk for Psychiatric Disorders. Sci Rep. 2018 Jul 30;8(1):11402. doi: 10.1038/s41598-018-29348-z. PMID 30061722
- [Background] Constantino DB, Xavier NB, Levandovski R, Roenneberg T, Hidalgo MP, Pilz LK. Relationship Between Circadian Strain, Light Exposure, and Body Mass Index in Rural and Urban Quilombola Communities. Front Physiol. 2022 Jan 26;12:773969. doi: 10.3389/fphys.2021.773969. eCollection 2021. PMID 35153809
- [Background] Pilz LK, Xavier NB, Levandovski R, Oliveira MAB, Tonon AC, Constantino DB, Machado V, Roenneberg T, Hidalgo MP. Circadian Strain, Light Exposure, and Depressive Symptoms in Rural Communities of Southern Brazil. Front Netw Physiol. 2022 Jan 26;1:779136. doi: 10.3389/fnetp.2021.779136. eCollection 2021. PMID 36925579
- [Background] Pilz LK, de Oliveira MAB, Steibel EG, Policarpo LM, Carissimi A, Carvalho FG, Constantino DB, Tonon AC, Xavier NB, da Rosa Righi R, Hidalgo MP. Development and testing of methods for detecting off-wrist in actimetry recordings. Sleep. 2022 Aug 11;45(8):zsac118. doi: 10.1093/sleep/zsac118. PMID 35598321
- [Background] Comiran Tonon A, Pilz LK, Amando GR, Constantino DB, Boff Borges R, Caye A, Rohrsetzer F, Souza L, Fisher HL, Kohrt BA, Mondelli V, Kieling C, Idiart M, Diez-Noguera A, Hidalgo MP. Handling missing data in rest-activity time series measured by actimetry. Chronobiol Int. 2022 Jul;39(7):964-975. doi: 10.1080/07420528.2022.2051714. Epub 2022 Mar 30. PMID 35350931
- [Background] Levandovski R, Dantas G, Fernandes LC, Caumo W, Torres I, Roenneberg T, Hidalgo MP, Allebrandt KV. Depression scores associate with chronotype and social jetlag in a rural population. Chronobiol Int. 2011 Nov;28(9):771-8. doi: 10.3109/07420528.2011.602445. Epub 2011 Sep 6. PMID 21895489
- [Background] Allebrandt KV, Teder-Laving M, Cusumano P, Frishman G, Levandovski R, Ruepp A, Hidalgo MPL, Costa R, Metspalu A, Roenneberg T, De Pitta C. Identifying pathways modulating sleep duration: from genomics to transcriptomics. Sci Rep. 2017 Jul 4;7(1):4555. doi: 10.1038/s41598-017-04027-7. PMID 28676676
- [Background] Alves Braga de Oliveira M, de Mendonca Filho EJ, Carissimi A, Lima Dos Santos Garay L, Scop M, Ruschel Bandeira D, Gutierrez Carvalho F, Mathur S, Epifano K, Adan A, Frey BN, Hidalgo MP. The Revised Mood Rhythm Instrument: A Large Multicultural Psychometric Study. J Clin Med. 2021 Jan 20;10(3):388. doi: 10.3390/jcm10030388. PMID 33498431
- [Background] Wittenbrink N, Ananthasubramaniam B, Munch M, Koller B, Maier B, Weschke C, Bes F, de Zeeuw J, Nowozin C, Wahnschaffe A, Wisniewski S, Zaleska M, Bartok O, Ashwal-Fluss R, Lammert H, Herzel H, Hummel M, Kadener S, Kunz D, Kramer A. High-accuracy determination of internal circadian time from a single blood sample. J Clin Invest. 2018 Aug 31;128(9):3826-3839. doi: 10.1172/JCI120874. Epub 2018 Aug 6. PMID 29953415